CLINICAL TRIAL: NCT05857410
Title: Clinical Effect Observation of Lower Limb Warming Blanket Combined With Dexmedetomidine in Preventing Postoperative Delirium and Chills in Elderly Patients Undergoing Spinal Surgery
Brief Title: Scheme of Limb Warming Blanket Combined With Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jincheng General Hospital (Other)
Responsible Party: Principal Investigator, Wei Fan, Principal Investigator, Jincheng General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: JinchengGH001
Record Dates: First submitted 2023-04-23; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Spine Surgery; Postoperative Delirium and Chills
Keywords: Elderly spinal surgery; Delirium and chills
MeSH Terms: conditions — Emergence Delirium; Chills; Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (group N) (No Intervention)
- heating group (group T) (Active Comparator)
  Interventions: Device: Lower limb heating blanket
- DEX group (group D) (Active Comparator)
  Interventions: Drug: Dexmetomidine
- heating combined with DEX group (group TD) (Experimental)
  Interventions: Drug: Dexmetomidine; Device: Lower limb heating blanket

INTERVENTIONS:
Drug: Dexmetomidine — Dexmetomidine (H20183219) 0.4μg / (kg·min)；
  Arms: DEX group (group D); heating combined with DEX group (group TD)
Device: Lower limb heating blanket — Beijing Maikang Medical Device Co., Ltd., Model: Warm-1-1.
  Arms: heating combined with DEX group (group TD); heating group (group T)

SUMMARY:
Objective: To observe the clinical effect of lower limb warming blanket combined with dexmedetomidine (DEX) in preventing postoperative delirium (POD) and chills in elderly patients undergoing spinal surgery. Methods: A total of 160 elderly patients undergoing posterior spinal surgery under general anesthesia were selected and divided into control group (group N), heating group (group T), DEX group (group D) and heating combined with DEX group (group TD) according to the random number table method, 40 cases in each group. T group and TD group routine insulation and lower limb heating blanket. DEX was injected in group D and group TD. The dosage of anesthetics, the changes of body temperature and heart rate at different time points during operation, and the occurrence of postoperative chills and POD were compared among the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 65-80 years old;
* American Society of Anesthesiologists (ASA) grade II-III;
* Normal body temperature before operation;
* the operation time was 2-4 hours

Exclusion Criteria:

* Preoperative fever or hypothermia (body temperature≥37.5 ℃ or≤35.5℃ on the day of operation);
* Body mass index (BMI) >30 kg/m2;
* The existence of heart, brain, lung, kidney and other important organs and circulatory system, respiratory system, immune system, central nervous system diseases;
* Patients who had taken antipsychotic drugs or β-blockers before surgery would have a greater impact on intraoperative body temperature and other patients who could not effectively cooperate with this study;
* Patients with operation time more than 5 hours

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Intraoperative vital signs monitoring | 1 hour
  nasopharyngeal temperature
Intraoperative vital signs monitoring | 2 hour
  nasopharyngeal temperature
Intraoperative vital signs monitoring | 3 hour
  nasopharyngeal temperature
The incidence of postoperative chills | 1 hour
  chills refer to the Wrench classification criteria as follows : 0: no chills; grade 1: peripheral vascular contraction, vertical hair, but no muscle fibrillation; level 2: only one muscle group had muscle fibrillation; grade 3: muscle fibrillation in multiple groups; level 4: general tremor; ≥ 1 level was judged to have chills.
The incidence of POD after operation | 1 day
  The results of POD in each group were recorded, and the POD was evaluated by CAM-CR scale. The incidence of POD at 24,48 and 72 h after operation was compared among the groups
Postoperative extubation time | 1 hour
  The recovery time from the end of surgery to extubation was recorded.
Postoperative incision infection rate | 1 hour
  The incidence of postoperative incision infection was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Jincheng General Hospital, Jincheng, Shanxi, China